CLINICAL TRIAL: NCT04919707
Title: Evaluation of Head Kinematics, Force-strain Models, and Correlation of MRI Markers With Neurocognitive Testing in Youth Soccer Heading
Brief Title: Youth Soccer Header Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-0048; A536110 (Other: UW Madison); SMPH/ORTHO&REHAB/ORTHO (Other: UW Madison); Protocol Version 4/26/2021 (Other: UW Madison)
Record Dates: First submitted 2021-05-25; First posted 2021-06-09 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Brain Injuries
Keywords: soccer; concussion; sports injuries
MeSH Terms: conditions — Brain Injuries; Brain Concussion; Athletic Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older Adolescent Soccer Players (Experimental): 10 male, 10 female soccer players, grades 11-12, age 16-18 Neurocognitive measures, physical measures, header session, MRI
  Interventions: Behavioral: Header Session; Procedure: MRI Session
- Younger Adolescent Soccer Players (Experimental): 10 male, 10 female soccer players, grades 6-7, age 12-13 Neurocognitive measures, physical measures, header session, MRI
  Interventions: Behavioral: Header Session; Procedure: MRI Session

INTERVENTIONS:
Behavioral: Header Session — Participant fit with commercially available Storelli ExoShield Head Guard that has been fit with head impact sensors; participant completes a set of basic standing header tasks which mimic the types of purposeful heading anticipated to occur in actual play in soccer practice and games.
Procedure: MRI Session — Scanning will include high resolution T1w imaging for 3-dimensional structural analyses, DTI and resting-state MRI for assessment of structural and functional brain network connectivity, as well as susceptibility-weighted imaging and multicomponent relaxometry to assess for microhemorrhages and myelin damage.

SUMMARY:
This study aims to establish and validate age-based head kinematics, force-strain models and brain injury probability maps from sensor worn data during soccer heading tasks. 40 youth soccer players will be recruited from the Madison, WI area and can expect to be on study for 2 months.

DETAILED DESCRIPTION:
Despite the large popularity of soccer worldwide and in the US, the majority of research on sport-related head impacts has been concentrated in male American football players using head-impact measurement sensors in instrumented football helmets. The limited research in soccer players likewise has focused on males, particularly those playing at an elite level, such as collegiate or professional. Unfortunately there is a paucity of data on youth soccer athletes in regards to how these younger players actually head the ball and what forces they experience. Measurement of head impacts is essential to further understanding the potential risks associated with heading in youth soccer, and to further inform rule or policy changes that limit head impact exposure in these younger age groups.

Specific Aim: Establish and validate age-based head kinematics, force-strain models and brain injury probability maps from sensor worn data during soccer heading tasks.

In this study, age-and sex-specific force strain models will be validated using a study of soccer headers under controlled conditions. Youth soccer players in 6th-12th grade will be recruited to participate in a header training session while wearing motion sensor headbands. All children will undergo MRI scanning and baseline assessment of neurocognitive function, psychological health, and academic aptitude and performance. Participant-specific finite element models will be created from MRI scans, and principle tissue strains will be determined based on head motion profiles during soccer headers and compared between age- and sex-specific groups.

High fidelity head kinematics will be acquired during soccer headers under controlled conditions using a custom headband embedded with multi-axis motion sensors. MRI scans will be obtained in all participants, and individualized and population averaged (to reduce computational burden), whole brain tractographs will be created. New participants-specific finite element models will be generated using geometry-adaptive mesh morphing techniques to match the head morphology of each subject using a baseline FE head model (to reduce model development time). The linear and angular acceleration histories obtained from the pre- and post-training soccer heading tasks will be applied directly to the FE models to simulate the head motion of each participant. The principal strains will be determined for each heading task, and brain injury probability maps will be generated based on the resulting tissue strain. Brain injury risk will be assessed through the incorporation of a cellular injury criterion embedded into the finite element simulations, with smaller strains correlating with lower injury risk. Soccer header force-strain relationships will be compared between age groups, and pre-and post-training session. This analysis will provide insight into the effect of age and training on improving heading techniques and reducing the risk of injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-13 or 16-18 years
* Currently participating in organized interscholastic or club soccer
* No active musculoskeletal injury that limits full participation in soccer activities

Exclusion Criteria:

* 14-15 year old are not eligible
* History of prior concussion or other head injury
* History of prior cervical spine injury
* Potential participants who can not participate in the MRI scan will be excluded
* Pregnancy or possible pregnancy (one reason for MRI exclusion)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Force Strain Kinematic Model Development: Maximum Strain | up to 2 months
  High fidelity head kinematics will be acquired during soccer headers under controlled conditions using a custom headband embedded with multi-axis motion sensors. Soccer header force-strain relationships will be compared between age groups, and pre-and post-training session.
Force Strain Kinematic Model Development: Minimum Principle Strain | up to 2 months
  High fidelity head kinematics will be acquired during soccer headers under controlled conditions using a custom headband embedded with multi-axis motion sensors. Soccer header force-strain relationships will be compared between age groups, and pre-and post-training session.
Force Strain Kinematic Model Development: Maximum Axonal Strain | up to 2 months
  High fidelity head kinematics will be acquired during soccer headers under controlled conditions using a custom headband embedded with multi-axis motion sensors. Soccer header force-strain relationships will be compared between age groups, and pre-and post-training session.
Whole brain tractography (fiber tracking) created by MRI scans | up to 2 months
  Whole brain tractographs will be created from MRI scans using Diffusion Tensor Imaging.
Brain Injury Probability Map Development: Change in Tissue Strain | During the header task session, up to 2 months
  The principal strains will be determined for each heading task, and brain injury probability maps will be generated based on the resulting tissue strain. Brain injury risk will be assessed through the incorporation of a cellular injury criterion embedded into the finite element simulations, with smaller strains correlating with lower injury risk.

SECONDARY OUTCOMES:
BRIEF-Monitoring Trail Making Parts A and B Score | up to 2 months
  The Trail Making Test is administered in two parts. Part A is a visual-scanning, timed task where subjects are asked to connect with lines 25 circles numbered from 1 to 25 as quickly as possible. In Part B participants are asked to connect circles containing numbers (from 1 to 13) or letters (from A to L) in an alternate numeric/alphabetical order (i.e. 1-A-2-B-3-C etc.). Errors must be corrected immediately and the sequence re-established. The TMT A-B score, calculated as the difference between TMT-A and TMT-B times, is considered a measure of cognitive flexibility relatively independent of manual dexterity.
Sport Concussion Assessment Tool 5 (SCAT5) Symptom Severity Score | up to 2 months
  The SCAT5 contains a 22 item concussion symptom evaluation scale with score of 0-6 for each symptom and total score 0-132, higher scores indicate more severe symptoms.
Sport Concussion Assessment Tool 5 (SCAT5) Number of Symptoms | up to 2 months
  The SCAT5 contains a 22 item concussion symptom evaluation scale with score of 0-6 for each symptom and total score 0-132, higher scores indicate more severe symptoms.
Patient Health Questionnaire (PHQ-9) Score | up to 2 months
  The PHQ-9 has 9 items with 0-3 scale for 0-27 total score. Higher score indicates greater level of depression. Scores of 0-4, 5-9, 10-14, 15-19 and >20 correspond to minimal or none, mild, moderate, moderately severe symptoms.
General Anxiety Disorder Scale-7 (GAD-7) Score | up to 2 months
  The GAD-7 has 7 items with 0-3 scale for 0-21 total score. Higher score indicates greater level of anxiety. Scores of 0-4, 5-9, 10-14, and 15-21 correspond to minimal or none, mild, moderate, and severe symptoms.
Pediatric Quality of Life Inventory (PEDS-QL) Score | up to 2 months
  The PedsQL is a generic measure of Health-related Quality of Life. The PedsQL consists of 23 questions that measure the domains of emotional, physical, social, and school function to calculate a physical and psychosocial summary as well as total score. The total score (23 items) is a summary score of all subscale scores (total range of scores from 0-92, higher scores indicate poorer quality of life), and the psychosocial functioning score (15 items) is a summary score of the emotional-functioning (5 items), social-functioning (5 items), and school-functioning (5 items) subscale scores (total range of scores from 0-60 where higher scores indicate poorer quality of life).
Deep Cervical Flexor Endurance Test (DCFET) | up to 2 months
  The subject lies supine flat on their back, tuck their chin toward their chest and lift their head and neck approximately 2.5 cm off the ground and hold that position as long as possible. The length of time is recorded in seconds, and typically is 45-60 sec.
Y Balance Test (YBT) | up to 2 months
  Leg length is measured (cm). The test consists of a centralized stance platform and three pipes connected with the platform. The pipes represent AT (Anterior), PM (Posterior Medial), and PL (Posterior Lateral) reach directions and are marked in 1.0-cm increments for measurement purposes. All pipes are equipped with a moveable reach indicator. During the testing procedure, subjects stand with one leg on the centralized platform and are instructed to reach with the other leg as far as possible in the AT, PM, and PL directions while maintaining balance. Each subject will perform three practice trials followed by three data collection trials per leg. Starting with the AT reach direction while standing on the right leg followed by standing on the left leg, this protocol is then replicated for the PM and PL directions.

CONTACTS AND LOCATIONS:
Overall Officials: M Alison Brooks, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No